CLINICAL TRIAL: NCT04166539
Title: Risk of Dementia and Heart Failure in Total Joint Arthroplasty
Brief Title: Neurotoxicity and Cardiotoxicity in Total Joint Arthroplasty
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Hilal Maradit Kremers, Principal Investigator, Mayo Clinic
Other Study IDs: 19-001294; R01AG060920 (NIH); R01HL147155 (NIH)
Record Dates: First submitted 2019-11-07; First posted 2019-11-18 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Metallosis; Pain; Total Hip Replacement; Total Knee Replacement
Keywords: Revision Surgery; Hip; Knee; Metals; Metallosis; Toxicity
MeSH Terms: conditions — Pain | interventions — Surveys and Questionnaires; Interviews as Topic; Blood Specimen Collection; Magnetic Resonance Spectroscopy; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metallosis Patients: Patients who are being seen by surgeons for metal-related issues in the blood, pain, or revision surgery.
  Interventions: Behavioral: Questionnaires; Behavioral: Interviews; Other: Blood draw; Radiation: Magnetic Resonance Imaging; Diagnostic Test: Echocardiogram
- Control Group: Patients who have had total hip or knee arthroplasty no less than 5-10 years ago, who have no symptoms.
  Interventions: Behavioral: Questionnaires; Behavioral: Interviews; Other: Blood draw; Radiation: Magnetic Resonance Imaging; Diagnostic Test: Echocardiogram

INTERVENTIONS:
Behavioral: Questionnaires — You will be asked to complete a questionnaire about your family history of neurological diseases and current and past physical thinking activities.
Behavioral: Interviews — Behavioral and Memory interviews will take place with the patient.
Other: Blood draw — Have a sample of blood drawn (4.2-5 tablespoons) for clinical and research tests.
Radiation: Magnetic Resonance Imaging — Each MR examination takes about 45 minutes and does not require the use of needles, medication or contrast enhancement. You will lie on your back and enter the MR scanner for the study, during which time you will hear knocking noises. People with pacemakers, aneurysm clips, cochlear implants, or metal/foreign objects in their eyes are not permitted to undergo MR studies. We will review your implants and determine your eligibility.
  Other Names: MRI
Diagnostic Test: Echocardiogram — Each echocardiogram takes about 30 minutes. This test uses sound waves to look at your heart. The person doing the test will press on your chest with a machine to obtain the pictures. The pressure may be uncomfortable. The echocardiogram will involve an image enhancement agent infusion to obtain better images.

SUMMARY:
The purpose of this research is to understand whether patients who previously had total hip or total knee replacement experience memory, thinking or heart problems. This study will help us determine if and how often these problems occur.

DETAILED DESCRIPTION:
At your first visit you will be asked to do the following.

* Sign this informed consent document.
* Questionnaire: You will be asked to complete a questionnaire about your family history of neurological diseases and current and past physical thinking activities.
* Interview: The interview will be performed by the study coordinator who is a member of the research team. It will take about 20-30 minutes to complete. You will be asked to answer questions about your general health, surgeries, medications, and your memory and thinking skills.
* Memory Interview: You will have an evaluation of your memory and thinking skills. You will answer questions and perform tasks that evaluate various thinking abilities such as concentration, memory, reasoning, and learning.
* Blood draw: Have a sample of blood drawn (4.2-5 tablespoons) for clinical and research tests.
* Magnetic Resonance Imaging (MRI) of your brain (optional): If you agree to participate, you will be asked to have MR imaging of your brain.
* Echocardiogram: You will be asked to have an echocardiogram of your heart.
* Follow-up visit in 2-3 years: You will be asked to return to Mayo for your second study visit in 2-3 years. At this visit, you will be asked to complete the same memory and thinking tests described for the first visit. You will also be asked to repeat the echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing to sign consent
* Patients scheduled for revision surgery for osteolysis, aseptic loosening, or wear of TJA implants/ALTR.

OR

-MCSA (Mayo Clinic Study of Aging) patients with THA or TKA with at least 10 years since surgery.

Exclusion Criteria:

* History of dementia
* History of cardiomyopathy or heart failure
* Revision for infection or fracture
* Patient is pregnant
* Patient has medication patches on
* Patient has a pacemaker or defibrillator (ICD)
* Patient has a deep brain stimulator (DBS)
* Patient has a vagal neuro stimulator (VNS)
* Patient has any other kind of neuro stimulator
* Patient has aneurysm clips in their head
* Patient has a tissue expander
* Patient has had a gastrointestinal clip or pill camera inserted in the last 90 days
* Patient has an esophageal reflux management system (LINX)
* Patient has a cochlear (ear) or auditory implant
* Patient has any implanted device (electronic or not) with magnets
* Patient has an eye injury involving metal
* Patient has allergy to contrast or dye

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients to complete cardiology part of the study (questionnaires, blood test, echocardiogram).
  100 patients to complete cognitive part of the study (questionnaires, interviews, blood test, MRI).
  Patient groups may overlap.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Mild Cognitive Impairment | 1 year
  Cognitive impairment as assessed through interviews
Brain MRI findings | 1 year
  imaging
Left ventricular dysfunction | 1 year
  heart dysfunction as assessed using echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Maradit Kremers, MD, Principal Investigator — Principal Investigator
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials